CLINICAL TRIAL: NCT01173107
Title: A Pilot Study for PK/PD Parameter of Colchicine in Chronic Kidney Disease Patient.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Suhnggwon Kim, Seoul National University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Colchicine_2010_1
Record Dates: First submitted 2010-07-28; First posted 2010-07-30 (Estimated); Last update posted 2010-12-29 (Estimated); Status verified 2010-12

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Colchicine

ARMS (1):
- MDRD eGFR 10~50 ml/min/1.73m2 (Experimental)
  Interventions: Drug: colchicine

INTERVENTIONS:
Drug: colchicine — colchicine 1T tid

SUMMARY:
A pilot study for PK/PD parameter of colchicine in Chronic kidney disease patient.

ELIGIBILITY:
Inclusion Criteria:

* from 18yrs to 80yrs , man and women
* the patient who are taking colchicine
* On screening, the patient shows that MDRD GFR >= 10 ml/min and <= 50 ml/min
* the patient sign on the concent form

Exclusion Criteria:

* the patient have experience to take medication that have an effect on renal function
* At least, the average level of two separate blood pressure ( 2min interval ) shows that SBP <= 100 mmHg or >=160 mmHg and DBP <=60 mmHg >=100 mmHg, or Heart rate < 40 beats/min or > 90 beats/min
* pregnancy or anticipate pregnancy with 6 month
* hypersensitivity to colchicine
* acute hepatitis or the level of AST or ALT is over 2times of normal range or the level of bilirubin is over 2.0 mg/dL
* serum albumin < 3.5 mg/dL or > 5mg/dL
* urinary retension, prostatic hyperplasia
* the patient show gout attack on taking colchicine
* the patient who have gastro-intestinal disease ( ex, crohn's disease, acute or chronic pancreatitis, ulcer )or who have the surgical history of gastrointestine.
* the patient who should take Atazanavir, Amprenavir, Apreptant, clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, diltiazem, erythromycin, fluconazole, fosamprenavir, grapefruit juice, verapamil, cyclosporine, ranolazine
* the patient who had taken part in the other study within 3months
* the patient who had gotten blood transfusion
* pregnant, breast feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-12; Primary Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
serum colchicine level | 0,1,6 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea